CLINICAL TRIAL: NCT05220735
Title: Effects of Omega-3 Fatty Acid Supplementation on Fractional Iron Absorption in South African Women Living With Obesity: A Stable Iron Isotope Study
Brief Title: Omega-3 Fatty Acid Supplementation and Fractional Iron Absorption in Obese South African Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: North-West University, South Africa (Other)
Responsible Party: Principal Investigator, Isabelle Herter-Aeberli, Senior Scientist, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FeMEGA-3
Record Dates: First submitted 2022-01-06; First posted 2022-02-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Obesity
Keywords: Fractional iron absorption; Inflammation; Omega-3 fatty acids
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants will receive three fish oil capsules daily for 14 weeks, and fractional iron absorption from test meals provided without and with ascorbic acid will be determined at baseline and endpoint.
  Interventions: Dietary Supplement: Omega-3 long chain polyunsaturated fatty acids (n-3 LCPUFA)

INTERVENTIONS:
Dietary Supplement: Omega-3 long chain polyunsaturated fatty acids (n-3 LCPUFA) — 3 three fish oil capsules providing 2.1 g n-3 PUFA; 1.27 g Docosahexanoic acid (DHA) and 0.86 g Eicosapentanoic acid (EPA) capsules.
  The absorption study test meals will consist of white bread with butter and honey, 6mg of labeled iron as ferrous sulfate and 300 g of distilled water. The meal will be given on two days without and with ascorbic acid. The test meals without ascorbic acid will contain 6 mg 57Fe as ferrous sulfate whereas the meals containing ascorbic acid will contain 6 mg 58Fe as ferrous sulfate.

SUMMARY:
In South Africa the prevalence of obesity in women of reproductive age is high; these women also have a high risk for iron deficiency (ID). Obesity is associated with low-grade systemic inflammation, which was shown to increase the expression of hepcidin, leading to a reduction in duodenal iron absorption. Thus, alleviating the sub-clinical inflammation associated with obesity could improve iron absorption and status. Supplementation with n-3 long-chain polyunsaturated fatty acids (LCPUFA) has been shown to reduce inflammation in obese individuals. A stable iron isotope study will be performed to investigate the effect of n-3 LCPUFA supplementation on fractional iron absorption in obese South African women.

DETAILED DESCRIPTION:
Iron deficiency (ID) and iron-deficiency anaemia (IDA) remain a major public health problem in low- and middle-income countries (LMICs). Women of reproductive age are at high risk of developing ID due to loss of iron through menstruation. Furthermore, inadequate iron status at conception and during pregnancy can have detrimental effects on the developing offspring. In addition to ID, the prevalence of obesity is increasing globally, including in LMICs. South Africa is a country with a high prevalence of obesity, especially in women of reproductive age (36 %), and a persistent burden of ID despite a mandatory maize meal and wheat flour fortification programme. Obesity is a condition associated with low-grade systemic inflammation. Inflammation increases the expression of hepcidin, leading to a reduction in duodenal iron absorption. Previous studies have shown that iron absorption differs between normal weight and obese individuals, and that the enhancing effect of ascorbic acid on iron absorption is lower in obese subjects. A possible explanation is the different sites of action of ascorbic acid and hepcidin on the enterocytes: Ascorbic acid enhances iron transport into enterocytes at the luminal side (via divalent metal transporter-1), while hepcidin reduces iron absorption by ferroportin inhibition at the basolateral membrane of the enterocyte. Thus, in obese individuals, an intervention at the basolateral membrane of the enterocyte will be needed. Supplementation with n-3 long-chain polyunsaturated fatty acids (LCPUFA) has been shown to exert cardiometabolic benefits, and to reduce inflammation in obese individuals.

The aim of this study is to investigate the effect of n-3 LCPUFA supplementation on fractional iron absorption in obese South African women of reproductive age. As a secondary objective, this study will determine association between omega-3 fatty acid status, inflammation and iron status in obese South African women. The hypothesises are: 1) fractional iron absorption will increase following n-3 LCPUFA supplementation; 2) iron absorption will further increase in the presence of ascorbic acid following n-3 LCPUFA supplementation.

After screening, apparently healthy, non-anaemic, obese South African women of African descent, aged 18 to 35 years, with low-grade inflammation and a low n-3 LCPUFA status, will receive daily oral fish oil (2.1 g of n-3 LCPUFA) capsules for three months. Iron status indices, inflammatory markers, hepcidin and omega-3 fatty acid index will be assessed at screening. The same variables will be emasured again at baseline and endpoint, in addition to erythrocyte total phospholipid fatty acid composition. Iron absorption will be determined from test meals with and without ascorbic acid using the oral stable isotope method, before (baseline) and after (endpoint) supplementation with n-3 LCPUFA.

ELIGIBILITY:
Inclusion Criteria:

* Self-classified women from African descent and of reproductive age (18 - 35 years)
* BMI ≥ 28kg/m2 (indicating obesity)
* Midly- or non-anaemic (Hb ≥11 g/dl)
* Low n-3 LCPUFA status (RBC omega-3 index < 6%)
* Low grade systemic inflammation (HS-CRP ≥ 2 mg/l but ≤ 20 mg/l)
* Be able to read and understand English

Exclusion Criteria:

* Treated chronic disease or gastrointestinal disorders
* Regular use of medication (except oral contraceptives, others after approval by the investigator) and women receiving treatment for high blood pressure
* Current consumption of iron or n-3 LCPUFA or ascorbic acid-containing supplements other than the supplements provided (Participants will be asked to discontinue use three weeks prior to enrolment)
* Subject on a weight loss diet or planning to start a weight loss diet during the duration of the study
* Pregnancy or lactation
* Subjects who cannot be expected to comply with the study protocol
* Subjects who are smoking
* Difficulty drawing blood due to poor quality veins
* Individuals that have a fear of needles or suffer from vaso-vagal episodes when exposed to blood
* Subjects with fish allergies
* Participants who plan to start or stop the use of contraceptives in the following 4 months.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of reproductive age
Enrollment: 33 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption (%) | Change between baseline and 3 months (days 17 and 118)
  Fractional iron absorption will be assessed from labeled meals consumed without and with ascorbic acid, before and after intervention with n-3 LCPUFA.

SECONDARY OUTCOMES:
Haemoglobin (g/dL) | Screening, days 1 and 102
  Haemoglobin will be measured in whole blood to determine presence of anaemia.
Ferritin (µg/L ) | Screening, days 1 and 102
  Ferritin will be measured in plasma to determine the presence of iron deficiency.
Soluble transferrin receptor (mg/L) | Screening, days 1 and 102
  Soluble transferrin receptor will be measured in plasma to determine the presence of iron deficiency.
Hepcidin concentration | Screening, days 1 and 102
  Hepcidin, a major regulator of iron absorption and influenced by inflammation, will be measured in plasma.
C-reactive protein (mg/L) | Screening, days 1 and 102
  C-reactive protein will be measured in plasma to determine the presence of acute inflammation.
Alpha-1-acid glycoprotein (g/L) | Screening, days 1 and 102
  Alpha-1-acid glycoprotein will be measured in plasma to determine the presence of chronic inflammation.
Intestinal fatty acid-binding protein | Screening
  Intesinal fatty acid-binding protein will be measured in plasma as a marker of intestinal damage.
Omega-3 fatty acid index (%) | Screening
  Omega-3 fatty acid index, a measure of eicosapentanoic and docosahexanic acids will be measued in red blood cells.
Cytokines (pg/ml) | Screening, days 1 and 102
  Cytokines: Interleukin (IL) IL-1α, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, Interferon gamma and Tumor necrosis factor-beta will be measured in plasma as markers of inflammation.
Erythrocyte fatty acid composition | Days 1 and 102
  Fatty acid composition and status will be determined in erythrocyte phospholipids.
Lipid mediators (mol/mL or pmol/mL) | Days 1 and 102
  The following lipid mediators will be measured in plasma: 17-Hydroxydocosahexanoic acid, 5-, 8-, 11-, 12-, 15- and 18-Hydroxyeicosapentanoic acid (HEPE); 5-, 8-, 11-, 12- and 15-Hydroxyeicosatetraenoic acids (HETE); Prostaglandinds E2, E3 and D2; Protectin D1 and Resolvin D1 and E1.
Genetic variants in genes associated with fatty acid metabolism | Days 1 and 102
  Single nucleotide polymorphism (SNP) analyses of genes involved in fatty acid metabolism will be measured from stored buffy coat.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Excellence for Nutrition, North-West University, Potchefstroom, South Africa

REFERENCES:
- [Derived] Uyoga MA, Baumgartner J, Malan L, Lewies A, Zandberg L, Zeder C, Smuts CM, Herter-Aeberli I. Omega-3 Long-Chain Polyunsaturated Fatty Acid Supplementation Did Not Reduce Inflammation to Improve Iron Absorption in South African Women Living with Overweight or Obesity. J Nutr. 2025 Dec 26:101280. doi: 10.1016/j.tjnut.2025.101280. Online ahead of print. PMID 41456679